CLINICAL TRIAL: NCT00883649
Title: A Randomized, Parallel-Group, Placebo-Control, Double-Blind Trial Comparing the Efficacy and Safety of Nutritional Supplementation Containing Omega 3 Fatty Acids and Gamma Linoleic Acid, for Treatment of Keratoconjunctivitis Sicca in Post-Menopausal Females
Brief Title: Efficacy and Safety Study of Nutritional Supplements for Treatments of Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Eye Consultants (Other)
Collaborators: ScienceBased Health (Industry); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SBH2005-01
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: Keratoconjunctivitis Sicca; Dry Eyes; Post-menopausal
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Other: Inactive Capsule
- 2 (Active Comparator)
  Interventions: Dietary Supplement: Hydroeye

INTERVENTIONS:
Dietary Supplement: Hydroeye — 2 Capsules BID
  Arms: 2
Other: Inactive Capsule — 2 Capsules BID
  Arms: 1

SUMMARY:
The purpose of this study is to determine the effectiveness of a nutritional supplement in post-menopausal women age 40 or older with moderate to severe dry eyes. This study is being conducted to determine if signs and symptoms of dry eye will improve with the use of this nutritional supplement.

ELIGIBILITY:
Inclusion Criteria:

* Signature on the written informed consent form
* Patient motivation and willingness to cooperate with the investigator by following the required medication regimen
* Patient willingness and ability to return for all visits during the study
* Rapid tear film break up time of eight seconds or less in at least one eye AND/OR
* Signs of meibomian gland dysfunction (MGD) including at least grade one lid notching, or the presence of orifice pustules
* At least grade one fluorescein superficial punctate keratitis (SPK) in at least one corneal quadrant or at least grade one conjunctival lissamine green staining in at least one eye.
* Ocular Surface Disease Index score of sixteen or greater.
* Willing to discontinue use of any current dry eye treatment (except artificial tears) for four weeks prior to randomization, and during the course of the six month study
* Post-menopausal women aged 40 years old or above. Post menopause is defined as absence of menstrual period for at least one year, or surgical hysterectomy with bilateral oophorectomy no less than six months prior
* If using transdermal, vaginal or systemic estrogen, progesterone, or estrogen derivatives, must be on a stable dose for at least 90 days, and be planning on staying on same stable dose for duration of the study

Exclusion Criteria:

* Concurrent involvement in any other clinical trial involving an investigational drug or device
* Compromised cognitive ability which may be expected to interfere with study compliance
* Uncontrolled or poorly controlled systemic disease (e.g., hypertension, diabetes) or the presence of any significant illness (e.g., serious gastrointestinal, renal, hepatic, endocrine, pulmonary, cardiac, neurological disease, cancer, AIDS, or cerebral dysfunction) that could, in the judgment of the investigator, jeopardize subject safety or interfere with the interpretation of the results of the study
* Known hypersensitivity to any components of the study or procedural medication
* Anticipated contact lens wear during the study
* History of corneal transplant
* Active ocular infection, uveitis or non-KCS inflammation
* History of recurrent herpes keratitis or active disease within the last six months
* History of cataract surgery within 3 months prior to enrollment
* History of ocular surface surgery (i.e. refractive, lasik, pterygium) within 6 months prior to enrollment
* corneal disorder or abnormality that affects corneal sensitivity or normal spreading of the tear film [except superficial punctate keratitis (SPK)]
* Use of systemic cyclosporine within prior 3 months
* Initiation, discontinuation or change in dosage of antihistamines, cholinergic agents, beta-blocking agents, tricyclic or SSRI antidepressants, phenothiazines, or topical or systemic acne rosacea medications in two months prior to enrollment, or anticipated change in dosage during course of study
* Topical ophthalmic medications within prior 4 weeks, or anticipated use of same during the study (except artificial tears)
* Use of Coumadin or Plavix within prior 2 weeks, or anticipated use of same during study. Stable dosing of aspirin 325mg or 85 mg per day is permitted.
* Use of fish oil, borage, evening primrose, flaxseed or black current seed oil supplements in the past three months
* Routine, usual dietary intake of more than 12 ounces of cold water fatty fish (tuna, salmon, mackerel, sea bass, sardines or herring) per week
* Occlusion of the lacrimal puncta either surgically or with temporary collagen punctal plugs within one month prior to study, or anticipated use of same during study
* A patient condition or situation which, in the judgment of the investigator, may put the patient at a significant risk, may confound the study results, or may interfere with the patient's participation in the study

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Schirmer tear test | Screening, Week 4, Week 12, Week 24
Ocular Surface Disease Index | Screening, Week 4, Week 12, Week 24
Tear Breakup Time | Screening, Week 4, Week 12, Week 24
Corneal Staining with Fluorescein | Screening, Week 4, Week 12, Week 24
Impression Cytology | Screening, Week 12, Week 24
Conjunctival staining with lissamine | Screening, Week 4, Week 12, Week 24

SECONDARY OUTCOMES:
Corneal Topography | Screening, Week 4, Week 12, Week 24
Meibomian Gland Dysfunction | Screening, Week 4, Week 12, Week 24
Facial Expression Subjective Scale | Screening, Week 4, Week 12, Week 24
Frequency of Artificial Tear Usage | Screening, Week 4, Week 12, Week 24
HLA-DR Staining of Impression Cytology | Screening, Week 12, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: John D Sheppard, M.D., Principal Investigator — Virginia Eye Consultants; Stephen C Pflugfelder, M.D., Principal Investigator — Baylor College of Medicine; Joe Wakil, M.D., Study Chair — ScienceBased Health; Penelope Edwards, MPH, CNS, Study Chair — ScienceBased Health
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Virginia Eye Consultants, Norfolk, Virginia

REFERENCES:
- [Derived] Sheppard JD Jr, Singh R, McClellan AJ, Weikert MP, Scoper SV, Joly TJ, Whitley WO, Kakkar E, Pflugfelder SC. Long-term Supplementation With n-6 and n-3 PUFAs Improves Moderate-to-Severe Keratoconjunctivitis Sicca: A Randomized Double-Blind Clinical Trial. Cornea. 2013 Oct;32(10):1297-304. doi: 10.1097/ICO.0b013e318299549c. PMID 23884332